CLINICAL TRIAL: NCT05965037
Title: Multicenter Prospective Registry in Current Clinical Practice With the Non-compliant Coronary Angioplasty Balloon Catheter. The FLUYDO NC Post Market Clinical Follow-up Study
Brief Title: The FLUYDO NC Post Market Clinical Follow-up Study
Status: Completed | Type: Observational
Sponsor: Alvimedica (Industry)
Collaborators: CID S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: C32103
Record Dates: First submitted 2023-05-30; First posted 2023-07-28 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Coronary Disease; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FLUYDO NC percutaneous transluminal coronary angioplasty balloon catheter — The FLUYDO NC is a rapid exchange percutaneous transluminal non-compliant coronary angioplasty balloon catheter. It is a single use only medical device, non-implantable, non-pyrogenic and sterilized with ethylene oxide and CO2 mixture. The distal portion has a hydrophilic coating and consists of two lumens: one for balloon inflation and deflation, the other for guidewire advancement and retraction. The product is indicated for balloon dilatation of the stenotic portion of a coronary artery or bypass graft stenosis for the purpose of improving myocardial perfusion.

SUMMARY:
The aim of the present observational study is to collect clinical data on the medical device non-implantable medical device Fluydo NC: coronary angioplasty non-compliant balloon dilatation catheter in the daily use in a not selected population.

ELIGIBILITY:
Inclusion Criteria:

* Turkish citizen,
* ≥18 years of age,
* Has indication for percutaneous transluminal coronary angioplasty (PTCA),
* Has indication to treat obstructive lesions of a native coronary artery or aortocoronary bypass or needs post dilatation of coronary stent
* Fluydo NC using in the primary lesion treated during the procedure by the decision physician,
* Has signed and dated the informed consent.

Exclusion Criteria:

* Has a previous diagnosis of coronary artery spasm in the absence of a significant stenosis.
* Needs the device use in an unprotected left main coronary artery
* Device use has not consistent with Instructions for Use.
* Participating in another medical device or pharmaceutical clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients meeting the patient selection criteria, over 18 years old, eligible for a catheter with FLUYDO NC catheter.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Device success | immediately after interventional procedure
Successful inflation, achievement of appropriate diameter, and deflation of the balloon | immediately after interventional procedure
Decrease in the percent stenosis after balloon procedure | immediately after interventional procedure
No perforation, flow-limiting dissection or reduction in Thrombolysis in Myocardial Infarction (TIMI) flow grade | immediately after interventional procedure
No life-threatening arrhythmias (sustained ventricular tachycardia, ventricular fibrillation) | immediately after interventional procedure

SECONDARY OUTCOMES:
Procedural success: Measurement: Percentage of device success without major adverse cardiovascular events (MACE) (composite of all death, myocardial infarction (MI), and clinically indicated target lesion revascularization (CI-TLR)) | Discharge or 48 hours after index procedure, whichever happens first
Rate of Target Lesion Failure (TLF) Measurement: Percentage of a composite of cardiac death, target vessel myocardial infarction (TV-MI), and CI-TLR. | discharge or 48 hours after index procedure, whichever happens first

CONTACTS AND LOCATIONS:
Locations (1):
- Alvimedica, Istanbul, Turkey (Türkiye)